CLINICAL TRIAL: NCT03422484
Title: Developpemment of a Score to Assess Risk of Medication Errors in Internal Medecin Unit
Brief Title: SCORE of Medication Error in Internal Medecin Unit
Acronym: SCOREME
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0030
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-02

CONDITIONS: Patient Hospitalized in Internal Medicine Unit
Keywords: Internal medecine unit; Medication Error; Clinical Pharmacist; Medication reconciliation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with at least one medication error: People with at least one medication error at hospital admission
  Interventions: Other: Detection and correction of medication error at hospital admission
- People without medication error at hospital admission: People without medication error at hospital admission

INTERVENTIONS:
Other: Detection and correction of medication error at hospital admission — Detection and correction of medication error at hospital admission
  Groups: People with at least one medication error

SUMMARY:
Transfers between interfaces of care are recognized as a source of medication discrepancies, medication errors (MEs) and potentially adverse drug events. ME are very common at hospital and may have important clinical and economic consequences. The lack and loss of medication information and communication between health professionals at points of care transition may often lead to ME. According to the literature, up to two thirds of medication histories contain at least one error. Some studies have compared pharmaceutical team with physician or nurse on the detection of UMD or ME and have reported that pharmacists were one of the best health care providers to establish medication history. To improve medication safety and decrease MEs rate, several institutions have recommended to develop medication reconciliation at all transition points such as admission, transfer and discharge. Medication reconciliation is the process that compares a patient's medication order to all medications that the patient has been taking and should take at admission, transfer and discharge of hospitalization. Medication reconciliation programs led by pharmacists are effective to reduce medications discrepancies. However, studies evaluating the efficacy of medication reconciliation program are very heterogeneous in terms of populations, definitions and methodology. Thus, proportion of ME differs enormously between studies, ranging from under 10% to over 60% at admission of hospitalization. Elderly patients with their numerous comorbidities associated with polypharmacy, such as patients of internal medecin unit, are at high risk of ME and at risk of safety issues. However, medication reconciliation process is very time consuming with an average of 30 minutes by patient. Thereby, review of all inpatients within 24 hours of admissions is very difficult or impossible. Targeting "high-risk situation" and "high-risk patient" are crucial to detect ME before causing harm. Therefore, evaluating the risk of MEs and their potential consequences in specific population of internal medicine unit using a validated medication reconciliation process seems of utmost importance for internal medicine specialist clinical practice and the decrease of ME rate. Consequently, the aim of our study was to (i) evaluate the prevalence of ME in an internal medicine unit at admission of hospitalization, (ii) determine the type of medication involved and the potential clinical impact of ME and (iii) identify factors associated with a risk of ME and serious ME.

ELIGIBILITY:
Inclusion criteria:

- Patients aged above 18 years old, admitted to the department during the study period and hospitalized for at least 24 hours

Exclusion criteria:

- NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of patient hospitalized in internal medecine unit of Montpellier University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1957 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
number of medication error | 1 day
  number of medication error at hospital admission detected by clinical pharmacist during medication reconciliation process

SECONDARY OUTCOMES:
number of variable associated to the risk of ME | 1 day
  number of variable associated to the risk of ME detected by logistic regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Audurier Y, Roubille C, Manna F, Zerkowski L, Faucanie M, Macioce V, Castet-Nicolas A, Jalabert A, Villiet M, Fesler P, Lohan-Descamps L, Breuker C. Development and validation of a score to assess risk of medication errors detected during medication reconciliation process at admission in internal medicine unit: SCOREM study. Int J Clin Pract. 2021 Feb;75(2):e13663. doi: 10.1111/ijcp.13663. Epub 2020 Dec 14. PMID 32770845